CLINICAL TRIAL: NCT00708084
Title: A Single-blind, Randomized, Monocentric Phase II Trial to Explore the Safety and Rabies-neutralizing Activity of Combined Administration of CL184 and Rabies Vaccine Versus Human Rabies Immune Globulin Plus Rabies Vaccine in Simulated Rabies Post-exposure Prophylaxis in Children and Adolescents
Brief Title: Randomized Phase II Trial on Safety and Neutralizing Activity of CL184 and Rabies Vaccine Versus Human Rabies Immune Globulin (HRIG) and Rabies Vaccine in Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAB-M-A004
Record Dates: First submitted 2008-07-01; First posted 2008-07-02 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Rabies
Keywords: Rabies post-exposure prophylaxis; Monoclonal antibody
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): CL184 combined with rabies vaccination
  Interventions: Biological: CL184
- B (Active Comparator): HRIG combined with rabies vaccination
  Interventions: Biological: HRIG

INTERVENTIONS:
Biological: CL184 — CL184 20 IU/kg intramuscularly on Day 0; in conjunction with rabies vaccine on Days 0, 3, 7, 14, and 28
  Arms: A
Biological: HRIG — HRIG 20 IU/kg intramuscularly on Day 0; in conjunction with rabies vaccine on Days 0, 3, 7, 14, and 28
  Arms: B

SUMMARY:
The aim of this study is to evaluate the safety of the monoclonal antibody cocktail CL184 in combination with rabies vaccine compared with human rabies immune globulin (HRIG) in combination with rabies vaccine in healthy children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Subjects free of obvious health-problems or with stable conditions
* Male or female subject aged ≥5 to ≤18 years
* Subject is living, studying, or working close to the study referral site
* Parent or legal representative signed written informed consent; in addition for subjects ≥12 years: signed assent form

Exclusion Criteria:

* Prior history of rabies exposure or immunization (rabies vaccine and/or immune globulin)
* Acute infection or disease within the last 2 weeks
* History and/or family history of clinically significant immunodeficiency or auto-immune disease
* Any history of known or suspected anaphylaxis or hypersensitivity reaction
* Planned immunization with live vaccines during the next 3 months
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of investigational medicinal product

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 42 days

SECONDARY OUTCOMES:
Rabies virus neutralizing activity | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz P. Quiambao, MD, Principal Investigator — Research Institute for Tropical Medicine, Alabang, Muntinlupa, Metro Manila, Philippines
Locations (1):
- Research Institute for Tropical Medicine, Alabang, Muntinlupa, Metro Manila, Philippines